CLINICAL TRIAL: NCT07234864
Title: An Exploratory Randomised, Double-Blind, Placebo-Controlled Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ZE63-0302 in Participants With Type 2 Diabetes Mellitus
Brief Title: Study to Assess Safety, Tolerability, PK, and PD of Multiple Doses of ZE63-0302 Administrated Orally in T2DM Patients.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eilean Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ZE63-0302-0002
Record Dates: First submitted 2025-09-25; First posted 2025-11-19 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; menin-inhibitor; type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZE63-0302 treatment (Experimental): Oral capsules BID
  Interventions: Drug: ZE63-0302
- Placebo (Placebo Comparator): Oral capsules BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ZE63-0302 — Oral capsules BID
  Arms: ZE63-0302 treatment
Drug: Placebo — Oral capsules BID
  Arms: Placebo

SUMMARY:
A Phase 1b study to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of multiple doses of ZE63-0302 administrated orally in T2DM patients.

DETAILED DESCRIPTION:
This is an exploratory randomised, double-blind, placebo-controlled study to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of 4-week treatment with ZE63-0302 versus placebo in participants with T2DM managed with up to 3 antidiabetic agents (except for insulin). Evaluation of dose levels will be conducted in a sequential fashion with lower dose levels evaluated first in the sequence. In this study patients will be enrolled to receive BID of ZE63-0302 or Placebo under fasted condition.

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent before any study-related activities are performed and must be able to understand the full nature and purpose of the study, including possible risks and adverse effects.
2. Adult males and females, ≥18 to ≤65 years of age (inclusive) at screening.
3. Diagnosis of T2DM of at least 7 years at the time of screening.
4. Must be receiving treatment with up to 3 antidiabetic agents (except insulin) at a stable, optimal, or maximum tolerated dose for at least 3 months prior to screening and with no dose changes expected during the study.
5. Must have HbA1c ≥7.5% and ≤9.5% at the screening visit.
6. Must have BMI ≥ 22.5 and ≤38.5 kg/m2 at the screening visit, with stable (± 5%) body weight within the previous 3 months of screening.
7. Female volunteers:

   1. Must be of non-childbearing potential, i.e., surgically sterilised (hysterectomy, bilateral salpingectomy, bilateral oophorectomy) at least 6 weeks before the screening visit or postmenopausal (where postmenopausal is defined as no menses for 12 months without an alternative medical cause and a follicle stimulating hormone [FSH] level consistent with postmenopausal status, per local laboratory guidelines), or
   2. If of childbearing potential, must:

   i. Have a negative pregnancy test at the screening visit and on Day 1. ii. Agree not to attempt to become pregnant or donate ova from signing the informed consent form (ICF) until at least 33 days after the last dose of study drug.

   iii. Agree to use adequate contraception (defined as use of a condom by the male partner combined with use of a highly effective method of contraception) from one month prior to screening until at least 33 days after the last dose of study drug, if not exclusively in a same-sex relationship or abstinent as a committed lifestyle.
8. Male volunteers:

   1. Must agree not to donate sperm from signing the ICF until at least 93 days after the last dose of study drug.
   2. If engaging in sexual intercourse with a female partner who could become pregnant, must agree to use adequate contraception (defined as use of a condom combined with use of a highly effective method of contraception) from signing the ICF until at least 93 days after the last dose of study drug.
   3. If engaging in sexual intercourse with a female partner who is not of childbearing potential or a same-sex partner, must agree to use a condom from signing the ICF until at least 3 days after the last dose of study drug.
9. Have suitable venous access for blood sampling, as determined by the investigator (or delegate).
10. Willing and able to comply with all study assessments, including performing SMPG and completing a study diary, and adhere to the protocol schedule and restrictions.

Exclusion Criteria:

1. Diagnosis of diabetes other than T2DM (e.g., type 1 diabetes, latent autoimmune diabetes of adults, monogenic diabetes, gestational diabetes) or at least one of the following at screening:

   1. Fasting C-peptide <0.8 ng/mL
   2. Fasting insulin >50 µIU/mL
2. Treatment with insulin within 3 months prior to or during screening.
3. Severe hypoglycaemia (defined as the occurrence of neuroglycopenic symptoms requiring the assistance of another person for recovery), hypoglycaemia unawareness, diabetic ketoacidosis, or non-ketotic hyperosmolar state within 3 months of screening.
4. Use of weight loss agents (Section 21.2) or diet (hypocaloric diet), unless the diet or weight loss treatment (prescription, herbal, over-the-counter, or other) has been stopped at least 3 months prior to screening and the participant has had stable (± 5%) body weight within the previous 3 months of screening.
5. Chronic systemic corticosteroid use, defined as any daily dose >10 mg prednisone or equivalent, for more than 2 consecutive weeks within 3 months prior to or during screening.

   Note: Topical, inhaled, ocular, nasal, or other non-systemic corticosteroid use is allowed.
6. Any use of hepatotoxic drugs (e.g., statins), gastric acid reducing medications, medications metabolized via the cytochrome P450 system (e.g., P-gp inhibitors, antifungal agents [ketoconazole, itraconazole], macrolides [erythromycin, clarithromycin], calcium channel blockers [verapamil, diltiazem], or medications with the potential for drug-drug interactions) within 3 months of screening.
7. Personal or family history (first-degree relative) of multiple endocrine neoplasia type 1.
8. History of or current acute or chronic pancreatitis or pancreatectomy.
9. History of or current liver cirrhosis, liver transplant, or any other liver disease including, but not limited to, the following: alcoholic liver disease, autoimmune or viral hepatitis, primary biliary cholangitis, primary sclerosing cholangitis, drug-induced hepatotoxicity, Wilson disease, clinically significant iron overload, or alpha-1-antitryspin deficiency requiring treatment.

   Note: Metabolic dysfunction-associated liver disease/metabolic dysfunction associated steatohepatitis without portal hypertension or cirrhosis and with acceptable liver function test results, as determined by the investigator (or delegate), is not exclusionary.
10. Significant inflammatory bowel disease, gastroparesis, or other severe disease or surgery affecting the gastrointestinal tract (including weight-reducing surgery and procedures) that could affect the interpretation of study data, as determined by the Investigator (or delegate).

    Note: Appendectomy, hernia repair, cholecystectomy, and similar conditions, as determined by the investigator (or delegate), are not exclusionary.
11. Any of the following events or conditions within 3 months prior to or during screening: hospitalisation due to unstable angina, myocardial infarction, coronary artery bypass graft or percutaneous transluminal coronary angioplasty, transient ischemic attack or significant cerebrovascular disease, or symptomatic heart failure (New York Heart Association Class III or IV).
12. Mean QT interval corrected using the Fridericia method (QTcF) >450 msec for men and >470 msec for women on screening ECG; or unstable, uncontrolled, or life-threatening arrhythmia or heart block, as assessed by the investigator (or delegate).
13. Untreated or unstable hypertension, defined as systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg after 10 minutes of supine rest and confirmed by repeated measurement at screening. Individuals with blood pressure above this threshold may have blood pressure-lowering medication(s) initiated and/or adjusted and be rescreened.
14. Any history of malignant disease in the last 5 years (excludes surgically resected squamous cell or basal cell carcinoma of the skin and cervical cancer in situ that have been treated with potentially curative therapy).
15. History of or current haemoglobinopathy (e.g., sickle cell anaemia, thalassaemia major, sideroblastic anaemia) or any other clinically important haematological abnormality (e.g., leucopoenia, thrombocytopaenia) as judged by the investigator (or delegate).
16. History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, haematological, gastrointestinal, endocrine, immunologic, dermatologic, psychiatric, or neurological disease/disorder, including any acute illness, within the past 3 months of screening, as determined by the investigator (or delegate) to be clinically relevant.
17. Any of the following laboratory abnormalities at screening:

    1. Aspartate aminotransferase ≥1.5 × upper limit of normal range (ULN)
    2. Alanine aminotransferase ≥1.5 × ULN
    3. Alkaline phosphatase (ALP) ≥1.5 × ULN
    4. Total bilirubin ≥1.5 × ULN (except for Gilbert's syndrome, which is not exclusionary, provided that direct (conjugated) bilirubin is ≤ ULN)
    5. Haemoglobin <11.5 g/dL (115 g/L) for males and <10.5 g/dL (105 g/L) for females
    6. Estimated glomerular filtration rate ≤60 mL/minute/1.73 m2 as defined by the Chronic Kidney Disease Epidemiology Collaboration formula
    7. Fasting triglycerides >400 mg/dL at screening Note: Individuals who fail screening based on this criterion must have their fasting status verified by the investigator (or delegate) and may have triglyceride-lowering medications adjusted and be retested during the screening window.
    8. Lipase and/or amylase ≥1.5 × ULN
    9. Thyroid stimulating hormone >6 mIU/L Note: Laboratory abnormalities (except for any exclusionary liver function test result) can be repeated once during the screening window at the discretion of the investigator (or delegate), if there is reasonable belief that the exclusionary result was obtained in error or is transient.
18. A history of or positive test results for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibodies at the screening visit.
19. Known or suspected history of alcohol or drug abuse within the past 3 years as judged by the investigator (or delegate).

    Note: Individuals on stable methadone or buprenorphine maintenance treatment for at least 12 months prior to screening may be included in the study.
20. Binge drinking behaviour or significant alcohol consumption, defined as consumption of >21 units/week if male and >14 units/week if female for a period of more than 3 consecutive months within 1 year prior to screening.
21. Known hypersensitivity to any of the proposed study treatments or ingredients/excipients.
22. Females who are breastfeeding or planning to breastfeed.
23. Donation of blood or plasma of ≥450 mL or loss of whole blood of ≥450 mL within 60 days prior to Day 1, or receipt of a blood transfusion within 60 days of Day 1, that may interfere with HbA1c determination.
24. Use of any vaccinations within 30 days prior to screening.
25. Administration of any investigational drug or participation in another interventional clinical study of an investigational drug or investigational device within 30 days or 5 half-lives of the investigational drug (whichever is longer) prior to screening.

    Note: Participation in an observational research study is not exclusionary.
26. Individuals who are employees, or close relative of an employee, of the Sponsor, CRO, or the study site, regardless of the employee's role.
27. Unavailability for follow-up assessments (e.g., planned major surgery during the study, relocation for job or family reasons) or concern for willingness or ability to follow study procedures (e.g., inability to complete long OGTT study visits, variable work schedule, travel, or shift work)
28. Any other condition or prior therapy that, in the opinion of the PI (or delegate), would make the individual unsuitable for this study, including inability to cooperate fully with the requirements of the study protocol or likelihood of noncompliance with any study requirements, or would interfere with evaluation of the study drug, put the individual at risk, or affect the interpretation of the results of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of AE/SAE. | From dosing to Week 4.
  To assess the incidence of adverse events and serious adverse events.
Change from baseline throughout the study in the vital signs and physical examination findings. | From dosing to Week 4.
Change from baseline throughout the study in 12-lead electrocardiogram results | From dosing to Week 4
Change from baseline throughout the study in Clinical laboratory assessments. | From dosing to Week 4.

SECONDARY OUTCOMES:
Half-life (t1/2) of ZE63-0302 | PK samples will be collected 15 minutes prior to dosing with ZE63-0302/Placebo to Day 28 6 hours post-dose.
Plasma Cmax | PK samples will be collected within 15 minutes prior to dosing with ZE63-0302/Placebo to Day 28 6 hours post-dose
  ZE63-0302 peak plasma concentration
Time to maximum concentration. | PK samples will be collected within 15 minutes prior to dosing with ZE63-0302/Placebo to Day 28 6 hours post-dose.
  ZE63-0302 time to maximum concentration.
Area under the concentration time curve from time 0 to 12 hours | PK samples will be collected within 15 minutes prior to dosing with ZE63-0302/Placebo to Day 28 6 hours post-dose.
Area under the concentration time curve from time 0 to 6 hours | PK samples will be collected within 15 minutes prior to dosing with ZE63-0302/Placebo to Day 28 6 hours post-dose.
Trough plasma concentration | PK samples will be collected within 15 minutes prior to dosing with ZE63-0302/Placebo to Day 28 6 hours post-dose.
Accumulation ratio. | PK samples will be collected within 15 minutes prior to dosing with ZE63-0302/Placebo to Day 28 6 hours post-dose.

OTHER OUTCOMES:
Absolute and percent change from baseline in Haemoglobin A1c and Fasting blood glucose. | From dosing to Week 4
Absolute and percent change from baseline in Fasting insulin, fasting C peptide, fasting glucagon, fasting C peptide-to-glucose ratio, and fasting proinsulin to-insulin ratio | From dosing to Week 4
Percent change from baseline to Week 12 in the AUC0 2h of Glucose, Insulin, C peptide, Glucagon, Incretin after OGTT. | From dosing to Week 4
Change from baseline in total cholesterol, high density lipoprotein, low density lipoprotein, triglycerides, and free fatty acids | From dosing to Week 4
Change from baseline in body weight | From dosing to Week 4
Absolute and percent change from baseline in HOMA2-%B and HOMA2-IR. | From dosing to Week 4.
Percent change from baseline to Week 12 in Insulin AUC0-2h/glucose AUC0-2h and C-peptide AUC0-2h/glucose AUC0-2h after OGTT. | From dosing to Week 4.
Percent change from baseline to Week 12 in additional C peptide-to-glucose or insulin to glucose indices and additional hormonal and biochemical parameters at different OGTT time points and AUC intervals | From dosing to Week 4
Change from baseline in waist circumference | From dosing to Week 4

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (4):
  - Emeritus Research Sydney, Botany, New South Wales
  - Momentum Clinical Research Taringa, Brisbane, Queensland
  - Momentum Clinical Research Sunshine, Melbourne, Victoria
  - Emeritus Research Camberwell, Melbourne, Victoria
- The Republican Specialized Scientific and Prectical Medical Center of Endocrinology named after Academician Yo. Kh. Turakulov, Tashkent, Tashkent, Uzbekistan

IPD SHARING:
Plan to Share IPD: No